CLINICAL TRIAL: NCT05837364
Title: Risk of Atrial Fibrillation and Association With Other Diseases: Protocol of the Derivation and International External Validation of a Prediction Model Using Nationwide Population-based Electronic Health Records
Brief Title: Predicting Risk of Atrial Fibrillation and Association With Other Diseases
Acronym: FIND-AF
Status: Completed | Type: Observational
Sponsor: University of Leeds (Other)
Collaborators: British Heart Foundation (Other); Clalit Health Services (Other); Ben-Gurion University of the Negev (Other)
Responsible Party: Principal Investigator, Dr Christopher Gale, Professor of Cardiovascular Medicine, University of Leeds
Other Study IDs: 318197
Record Dates: First submitted 2023-04-18; First posted 2023-05-01 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Atrial Fibrillation; Arrhythmias, Cardiac; Heart Diseases; Cardiovascular Diseases; Pathologic Processes
Keywords: Computation; Data Science
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac; Heart Diseases; Cardiovascular Diseases; Pathologic Processes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Development of an algorithm — Development of an algorithm to predict the risk of new onset Atrial Fibrillation

SUMMARY:
Atrial fibrillation (AF) is a major public health issue: it is increasingly common, incurs substantial healthcare expenditure, and is associated with a range of adverse outcomes. There is rationale for the early diagnosis of AF, before the first complication occurs. Previous AF screening research is limited by low yields of new cases and strokes prevented in the screened populations. For AF screening to be clinically and cost-effective, the efficiency of identification of newly diagnosed AF needs to be improved and the intervention offered may have to extend beyond oral anticoagulation for stroke prophylaxis. Previous prediction models for incident AF have been limited by their data sources and methodologies. An accurate model that utilises existing routinely-collected data is needed to inform clinicians of patient-level risk of AF, inform national screening policy and highlight opportunities to improve patient outcomes from AF screening beyond that of only stroke prevention. The investigators will use routinely-collected hospital-linked primary care data to develop and validate a model for prediction of incident AF within a short prediction horizon, incorporating both a machine learning and traditional regression method. They will also investigate how atrial fibrillation risk is associated with other diseases and death. Using only clinical factors readily accessible in the community, the investigators will provide a method for the identification of individuals in the community who are at risk of AF, thus accelerating research assessing whether atrial fibrillation screening is clinically effective when targeted to high-risk individuals.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is a major public health issue: it is increasingly common, incurs substantial healthcare expenditure, and is associated with a range of adverse outcomes. There is rationale for the early diagnosis of AF, before the first complication occurs. Previous AF screening research is limited by low yields of new cases and strokes prevented in the screened populations. For AF screening to be clinically and cost-effective, the efficiency of identification of newly diagnosed AF needs to be improved and the intervention offered may have to extend beyond oral anticoagulation for stroke prophylaxis. Previous prediction models for incident AF have been limited by their data sources and methodologies. An accurate model that utilises existing routinely-collected data is needed to inform clinicians of patient-level risk of AF, inform national screening policy and highlight opportunities to improve patient outcomes from AF screening beyond that of only stroke prevention.

The application of Random Forest will be investigated and multivariable logistic regression to predict incident AF within a 6 months prediction horizon, that is a time-window consistent with conducting investigation for AF. The Clinical Practice Research Datalink (CPRD)-GOLD dataset will be used for derivation, and the Clalit Health Services dataset will be used for international external geographical validation. Both comprise a large representative population and include clinical outcomes across primary and secondary care. Analyses will include metrics of prediction performance and clinical utility. Only risk factors accessible in the community will be used and the model could thus enable passive screening for high-risk individuals in electronic health records that is updated with presentation of new data. The study aims to create a calculator from a parsimonious model. Kaplan-Meier plots for individuals identified as higher and lower predicted risk of AF will be calculated and derive the cumulative incidence rate for non-AF cardio-renal-metabolic diseases and death over the longer term to establish how predicted AF risk is associated with a range of new non-AF disease states.

To ascertain whether the prediction model is transportable to geographies outside of the UK, the model's performance will be externally validated in the Clalit Health Services database in Israel. The validation will include participants insured by Clalit with continuous membership for at least 1 year before 01/01/2019: 2,159,663 patients with 4,330 of them having a new incident of AF (Atrial fibrillation and/or atrial flutter) in the first half of 2019. The study population will comprise all available patients who have at least 1-year follow up. The outcome of interest is the first diagnosed AF after baseline and will be identified using Read codes and ICD-9/10 codes. Patients with less than one year of registration, who are under thirty years of age at point of study entry, or have a preceding diagnosis of atrial fibrillation, will be excluded.

ELIGIBILITY:
Inclusion Criteria:

A least 1 year follow-up

Exclusion Criteria:

Diagnosed AF before study entry

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The derivation dataset will be the Clinical Practice Research Datalink-GOLD (CPRD-GOLD) dataset. The extracted dataset, including linked data, comprises all patients for the period between 2nd January 1998 and 30th November 2018 from the snapshot of CPRD-GOLD in October 2019.
Sampling Method: Non-Probability Sample
Enrollment: 2159663 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
1. To develop and validate a model for predicting the risk of new onset AF within the next 6 months | Between 1st Jan 1998 and 31st December 2018
  a. Predictive factors will be identified using Read codes and ICD-9/10 codes (diagnoses) Variables considered as potential predictors may include sociodemographic variables (age, sex, ethnicity) and morbidities.
1. To quantify the association between risk of new-onset AF and the hazard of other cardio-renal-metabolic diseases and death | Between 1st Jan 1998 and 31st December 2018
  a. All patients categorized as lower or higher predicted AF risk by the developed prediction model will be included. The initial presentation of a cardiovascular, renal, or metabolic disease or death will be considered because AF is associated with a high risk of adverse clinical outcomes. The occurrence of death by any cause will be quantified. Incident diagnoses will be defined as the first record of that condition in primary or secondary care records from any diagnostic position. Kaplan-Meier plots will be created for individuals identified as higher and lower predicted risk of AF and derive the cumulative incidence rate for each outcome at 1, 5 and 10 years considering the competing risk of death, as well as death at 5 and 10 years. For each specified outcome, the hazard ratio (HR) will be calculated between higher and lower predicted risk of AF using the Fine and Gray's model with adjustment for the competing risk of death.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher P Gale, Principal Investigator — University of Leeds
Locations (1):
- University of Leeds, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared.

REFERENCES:
- [Derived] Nadarajah R, Wu J, Arbel R, Haim M, Zahger D, Benita TR, Rokach L, Cowan JC, Gale CP. Risk of atrial fibrillation and association with other diseases: protocol of the derivation and international external validation of a prediction model using nationwide population-based electronic health records. BMJ Open. 2023 Dec 9;13(12):e075196. doi: 10.1136/bmjopen-2023-075196. PMID 38070890